CLINICAL TRIAL: NCT01140191
Title: An Open-Label Clinical Study to Examine the Safety, Efficacy, and Pharmacokinetics of WR 279,396 (Paromomycin + Gentamicin Topical Cream) for the Treatment of Cutaneous Leishmaniasis at Walter Reed National Military Medical Center (WRNMMC)
Brief Title: Safety, Efficacy, and PK of Topical Paromomycin/Gentamicin Cream for Treatment of Cutaneous Leishmaniasis
Acronym: WRNMMC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was closed due to lack of enrollment (only one subject enrolled)
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-16049; S-10-0007; USAMMDA Protocol Number (Other: PG-WRAMC-08-01)
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: leishmaniasis; cutaneous; WR 279,396; paromomycin; gentamicin; pharmacokinetics; safety; efficacy; military
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WR 279,396 (Experimental): All subjects in this one-arm study will receive topical WR 279,396
  Interventions: Drug: WR 279,396

INTERVENTIONS:
Drug: WR 279,396 — Topical application of WR 279,396 cream (15% paromomycin + 0.5% gentamicin)once daily for 20 days
  Other Names: Topical Paromomycin/Gentamicin Cream

SUMMARY:
The objectives of the study are to evaluate the safety, pharmacokinetics (PK), and efficacy of open label treatment with WR 279,396 (Topical Paromomycin/Gentamicin Cream)in subjects with cutaneous leishmaniasis (CL).

DETAILED DESCRIPTION:
Subjects will be screened over a period of up to 14 days prior to first treatment, and will receive treatment once daily for 20 days. Safety will be assessed by monitoring AEs, lesion site reactions, vital signs, hematology, and blood chemistry parameters.

Complete cure of ulcerated lesions is defined as 100% re-epithelialization or a measurement of ulceration of 0 x 0 mm. non-ulcerated treated lesions will also be measured to monitor total area of exposure of lesions to study drug and will be evaluated for cure (the absence of raised area on the skin).

Follow-up evaluations will be at 28 +2 days, 60 +7 days and 100 +14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female military health care beneficiary of any race or ethnicity and at least 18 years of age
* Subjects must give written informed consent.
* Subjects must have a diagnosis of CL in at least one lesion by at least one of the following methods: 1) positive culture for promastigotes; 2) microscopic identification of amastigotes in stained lesion tissue; 3) positive polymerase chain reaction (PCR) assay; and/or 4) prior diagnosis of CL within 14 days of the start of treatment.
* Subjects must have at least one ulcerative lesion ≥ 1 cm and < 5 cm, that meets the criteria for an index lesion (Larger lesions will be accepted for treatment, but these will not be included in the primary evaluation of efficacy).
* Subjects must be willing to forego other forms of treatments for CL including other investigational treatment during the study.
* Subjects must be capable of understanding and complying with the protocol (in the opinion of the investigator).
* Subjects must expect to be located in the Washington DC metropolitan area for at least the duration of the screening, 20-day treatment period, and Day 28 +/- 2 days follow-up visit.
* Subjects who are female and of child-bearing potential, must have a negative pregnancy test during screening and agree to use an acceptable method of birth control during the treatment phase and for 1 month after treatment is completed.
* Subject has adequate venous access for blood draws, if consented to the PK part of study.

Exclusion Criteria:

* Subject has had a prior diagnosis of leishmaniasis where all lesions had healed.
* Subject has only a single lesion whose characteristics include any of the following: verrucous or nodular lesion (non-ulcerative), lesion <1 cm in its greatest diameter, lesion in a location that in the opinion of the Investigator is difficult to maintain application of study drug topically.
* Subject has a lesion due to Leishmania that involves the mucosa or palate.
* Subject has signs and symptoms of disseminated disease.
* Subject is a female who is breast-feeding.
* Subject has an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed.
* Subject has significant organ abnormality, chronic disease such as diabetes, severe hearing loss, evidence of renal or hepatic dysfunction, or creatinine, AST, or ALT greater than the upper limit of normal as defined by the clinical laboratory normal ranges.
* Subject has received treatment for leishmaniasis including thermosurgery (ThermoMed™) or any medication with pentavalent antimony including sodium stibogluconate (Pentostam), meglumine antimoniate (Glucantime); amphotericin B (including liposomal amphotericin B and amphotericin B deoxycholate); WR 279,396; or other medications containing paromomycin (administered parenterally or topically) or methylbenzethonium chloride (MBCL); gentamicin; fluconazole; ketoconazole; pentamidine; or allopurinol within 4 weeks of starting study treatment.
* Subject has a history of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides.
* Subject has any other topical disease/condition which interferes with the objectives of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whitman, DO, USN, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was held 06Sep13 thru 17Dec2013 at study center WRNMMC at Bethesda 8901 Wisconsin Ave., Building 7, 1st Floor Bethesda, MD 20889
Pre-assignment Details: Statistical analysis was not performed as only a single subject was enrolled. No PK analysis was performed as this subject elected not to participate in the PK part of the study.
Period: Overall Study
Arm/Group | WR 279,396
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only 1 patient enrolled
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
Number of Lesions [Number; unit: Lesions] | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Application site reactions including elicited question about pain, and clinician examination for erythema/redness and swelling/edema Blood chemistries and hematology Vital signs
Time Frame: 3 months
Population: Analysis was per protocol
Measure: Number; unit: Adverse Events
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Adverse Events | 3

2. Primary Outcome: 100% Re-epithelialization of Index Lesion by Nominal Day 60
Description: Number of participants with 100% re-epithelialization of index lesion by nominal Day 60
Time Frame: Day 60
Population: Analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: Number of Participants Demonstrating Initial Clinical Improvements
Description: Number of participants with > 50% re-epithelialization of index lesion by Day 60 followed by complete re-epithelialization of index lesion on or before nominal Day 100;
Time Frame: 60-100 days
Population: Analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Participants | 1

4. Primary Outcome: Number of Participants With No Relapse of Index Lesion Between Nominal Day 60 and 100
Description: Number of participants with no relapses of lesion between 60 and 100 days. Relapse is defined as a 10% or greater increase in the area of ulceration of the index lesion or a shift from 100% re-epithelialization to < 100% re-epithelialization of the index lesion at Day 100 for those subjects that had 100% re-epithelialization of the index lesion at nominal Day 60 or before
Time Frame: 60-100 days
Population: Analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Cures of All Other Lesions
Description: Number of participants with 100% re-epithelialization of all ulcerated lesions and resolution of all other types of lesions
Time Frame: 100 days
Population: Analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Complete Cure of Index Lesion by Day 100
Description: Number of participants with complete cure of index lesion by day 100. Cure rate is defined as 100% re-epithelialization of an ulcerated lesion
Time Frame: 100 days
Population: Analysis per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 100 days
Description: Duration of treatment was 20 days, total days for event reporting was 100.
Arm/Group | WR 279,396
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WR 279,396 (N=1)
Headache (Nervous system disorders) | 1 (1) — Moderate in severity with an unlikely relationship to study. No action was taken and issue resolved
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) — Moderate in severity. Unlikely related to study. No action was taken and issue resloved
Application Site Pruritus (General disorders) | 1 (1) — Mild in severity. Probably related to study. No action was taken and issue resolved.

LIMITATIONS AND CAVEATS:
Only one subject was enrolled in the protocol and treated. Data for this single patient was the only data available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No